CLINICAL TRIAL: NCT07177781
Title: Longer-term Effects of Wild Blueberry Consumption on Brain Function in Older Men and Women
Brief Title: Effects of Wild Blueberry Consumption on Brain Function in Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Wild Blueberry Association of North America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 24-040
Record Dates: First submitted 2024-11-12; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2024-11

CONDITIONS: Brain Insulin-sensitivity; Brain Vascular Function; Cerebral Blood Flow
Keywords: Cognitive performance; Brain insulin-resistance; Brain vascular function; Cerebral blood flow; Wild blueberry; Brain insulin-sensitivity; Anthocyanin

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, controlled cross-over design. Participants will receive, in a random order, daily 26 grams of wild blueberry powder or a matched placebo for sixteen weeks, separated by a washout period of at least 8 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Matched placebo (No Intervention): Adults will receive in a random order, freeze-dried wild blueberry powder or a matched placebo for sixteen weeks, with a wash-out period of minimal eight weeks in-between. The placebo is an appearance, taste and macronutrient, fiber and vitamin C-matched powder containing blueberry flavoring and aroma, coloring, glucose, fructose, citric acid, ascorbic acid, cellulose, fibersol-2, xanthin gum, pectin, and silica. The placebo does not contain any form of anthocyanin that could potentially interfere with the wild blueberry intervention.
- Wild blueberry powder (wild blueberry intervention) (Experimental): The wild blueberry intervention consist of 100% freeze-dried wild blueberry powder, containing anthocyanins. Participants will consume daily 26 grams of freeze-dried wild blueberry powders for 16 weeks. Participants should consume the powders by mixing them with water once daily in the morning
  Interventions: Dietary Supplement: Wild blueberry powder

INTERVENTIONS:
Dietary Supplement: Wild blueberry powder — Study volunteers will consume daily 26 grams of wild blueberry powder for 16 weeks, which has to be dissolved in a glass of water.
  Arms: Wild blueberry powder (wild blueberry intervention)

SUMMARY:
Impaired brain vascular function precedes the development of reduced cognitive performance, while brain insulin-resistance is associated with cognitive decline. Evidence from epidemiological studies has already suggested beneficial effects of wild blueberry consumption on cognitive performance. However, underlying mechanisms have not yet been established, while well-controlled trials on longer-term effects of wild blueberries on cognitive performance are highly needed. This study hypothesizes that longer-term wild blueberry intake improves (regional) brain vascular function and insulin-sensitivity, thereby improving cognitive performance in older men and women. The primary objectives are to investigate in older adults the effect wild blueberry consumption on (regional) vascular function and insulin-sensitivity in the brain, and to focus on changes in cognitive performance as assessed with the CANTAB neuropsychological test battery (i.e., secondary objective). Cerebral blood flow responses before (brain vascular function) and after the administration of intranasal insulin spray (brain insulin-sensitivity) will be non-invasively quantified by the non-invasive gold standard magnetic resonance imaging (MRI)- perfusion method Arterial Spin Labeling (ASL).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged between 60-75 years
* BMI between 25-35 kg/m2 (overweight or obese)
* Fasting plasma glucose < 7.0 mmol/L
* Fasting serum total cholesterol < 8.0 mmol/L
* Fasting serum triacylglycerol < 4.5 mmol/L
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study.
* No difficult venipuncture as evidences during the screening visit.

Exclusion Criteria:

* Allergy or intolerance to berries
* Left-handedness
* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic consumptions per day
* Use of products or dietary supplements known to interfere with the main outcomes as judged by the principal investigators
* Use medication to treat blood pressure, lipid, or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases, and rheumatoid arthritis.
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident.
* Contra-indications for MRI imaging (e.g., pacemaker, surgical clips/material in body, metal splinter in eye, claustrophobia)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
MRI-brain perfusion measurement Arterial Spin Labeling | Change in brain perfusion at the end of a 16-week wild blueberry intervention and a 16-week control period with a matched placebo.
  Cerebral blood flow responses before (brain vascular function) and after the administration of intranasal insulin (brain insulin-sensitivity) will be non-invasively quantified by MRI-perfusion method Arterial Spin Labeling (ASL).

SECONDARY OUTCOMES:
Cognitive performance measurement by Cambridge Neuropsychological Test Automated Battery | Change in cognitive performance at the end of a 16-week wild blueberry intervention and a 16-week control period with a matched placebo.
  Cognitive performance will be investigated using Cambridge Neuropsychological Test Automated Battery (CANTAB), which will be performed on an Ipad. The cognitive task performance will be tested in three important cognitive domains namely attention, memory and executive function. Learning effects are prevented by randomization of the intervention periods and the settings of CANTAB, including parallel modes and stimuli randomization. The test will be performed in Dutch.
Brain Insulin Sensitivity | Change in outcomes at the end of a 16-week wild blueberry intervention and 16-week control period with a matched placebo.
  Change in cerebral blood flow, as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL), before and after application of intranasal insulin (160 IU).

OTHER OUTCOMES:
Assessment of Glucose Metabolism by 7-Point OGTT | Change in glucose metabolism at the end of a 16-week wild blueberry intervention and a 16-week control period with a matched placebo.
  Glucose metabolism will be evaluated using a 7-point oral glucose tolerance test (OGTT). In this test, a participant drinks a glucose-containing solution, and blood samples are collected at seven time points (0', 15', 30', 45', 60', 90', 120') over two hours. Measuring glucose levels at seven different points provides a detailed picture of how the body processes and clears sugar from the blood, helping to identify early changes in insulin sensitivity and overall metabolic health.
Assessment of cardiovascular function by Flow-Mediated Vasodilation (FMD) | Change in cardiovascular function at the end of a 16-week wild blueberry intervention and a 16-week control period with a matched placebo.
  Vascular health will be assessed by flow-mediated vasodilation (FMD, expressed as %), a non-invasive ultrasound technique that measures how well a blood vessel widens in response to increased blood flow. By briefly restricting blood flow in the arm (by means of a cuff on the fore arm) and then releasing it, investigators can see how effectively the brachial artery relaxes and dilates. This response reflects the function of the endothelium, the inner lining of blood vessels, and is considered an important indicator of cardiovascular health. The percentage indicates the relative increase in the brachial diameter compared to its baseline size.
Assessment of cardiovascular function by Carotid Artery Reactivity (CAR) | Change in peripheral vascular function at the end of a 16-week wild blueberry intervention and a 16-week control period with a matched placebo.
  The peripheral vascular function will be assessed by the carotid artery reactivity (CAR, expressed as %), a non-invasive technique that evaluates the ability of the carotid artery to dilate or constrict in response to specific physiological or pharmacological stimuli. The percentage indicates the relative change in the carotid artery's diameter compared to its baseline size. This method provides insight into endothelial function, vascular smooth muscle responsiveness, and overall arterial health, serving as an early marker for cardiovascular risk.
Assessment of Arterial Stiffness by Pulse Wave Analysis (PWA) | Change in arterial stiffness at the end of a 16-week wild blueberry intervention and a 16-week control period with a matched placebo.
  Arterial stiffness and central blood pressure will be assessed by pulse wave analysis (PWA). This non-invasive method records the shape of the pulse wave generated by each heartbeat, from the wrist or arm. From this signal, central blood pressure is expressed in millimeters of mercury (mmHg), while derived indices of arterial stiffness (such as the augmentation index, AIx) are expressed in percentages (%), representing the relative contribution of reflected waves to the overall pulse wave. By analyzing how the wave travels and reflects in the arteries, investigators can gain insight into arterial elasticity, vascular resistance, and the overall condition of the cardiovascular system.
Assessment of arterial stiffness by Pulse Wave Velocity (PWV) | Change in outcomes at the end of a 16-week wild blueberry intervention and a 16-week control period with a matched placebo.
  Arterial stiffness will be assessed by pulse wave velocity (PWV, expressed in meters per second [m/s]). This non-invasive technique measures the speed at which the pressure wave created by the heartbeat travels through the arteries. Since stiffer arteries allow the wave to move faster, PWV provides a reliable indicator of vascular elasticity and cardiovascular risk.
Assessment of microvasculature by Retinal Microvascular Calibers | Change in outcomes at the end of a 16-week wild blueberry intervention and a 16-week control period with a matched placebo.
  The microcirculation will be assessed by measuring retinal microvascular calibers. Using non-invasive retinal imaging, the diameters of small blood vessels in the back of the eye are quantified. Because the retina offers a unique 'window' to the body's microvascular system, changes in these tiny vessel widths can reveal early signs of vascular dysfunction and give an indication about cardiometabolic health.
Measuring blood pressure using office and 24-hour ambulatory monitoring | Change in outcomes at the end of a 16-week wild blueberry intervention and a 16-week control period with a matched placebo.
  Blood pressure (systolic and diastolic) and heart rate will be assessed through both office measurements and 24-hour ambulatory monitoring. Office blood pressure provides standardized readings taken in a clinical setting, while ambulatory blood pressure monitoring records values at regular intervals throughout the day (every 15 minutes) and night (every 30 minutes) as individuals go about their daily lives. Together, these methods give a more complete picture of blood pressure patterns, capturing variability, nighttime values, and potential masked or white-coat hypertension.
Assessment of blood lipids: TAG, TC, and HDL-C | Change in blood lipids at the end of a 16-week wild blueberry intervention and a 16-week control period with a matched placebo.
  Blood lipid levels will be assessed by measuring triacylglycerol (TAG), total cholesterol (TC), and high-density lipoprotein cholesterol (HDL-C). These standard blood tests provide important information about fat metabolism and cardiovascular risk.
Assessment of blood glucose levels | Change in blood glucose levels at the end of a 16-week wild blueberry powder and a 16-week control period with a matched placebo.
  Blood glucose will be measured from blood samples to determine the concentration of sugar in the bloodstream. Measuring blood glucose provides important information about metabolic health.
Evaluation of metabolic function by insulin measurement | Change in outcomes at the end of a 16-week wild blueberry intervention and 16-week control period with a matched placebo.
  Insulin levels will be measured from blood samples to evaluate how the body regulates glucose. Measuring insulin provides insight into metabolic function and insulin sensitivity.
Metabolic risk markers - Low-grade systemic inflammation | Change in metabolic risk markers at the end of a 16-week wild blueberry intervention and 16-week control period with a matched placebo.
  Markers for low-grade systemic inflammation (IL-6,TNF-alfa) will be assessed in the blood plasma to determine low-grade systemic inflammation.
High-resolution structural brain imaging with MPRAGE | Change in outcomes at the end of a 16-week wild blueberry intervention and 16-week control period with a matched placebo.
  Brain structure will be assessed using a structural MRI with an MPRAGE sequence. This high-resolution imaging technique provides detailed pictures of brain anatomy, allowing investigators to examine the size and shape of different brain regions.
Single nucleotide polymorphism (SNPs) | Change in outcomes at baseline measurements at the start of a 16-week wild blueberry intervention and a 16-week control period with a matched placebo.
  Leucocytes will be isolated from EDTA blood. DNA will be isolated from these leucocytes according to standard procedures. DNA will be used for analyzing the presence of known SNPs in genes encoding proteins known to play a role in cholesterol metabolism.
Other perceivable benefits: Assessment of Quality of Life | Change in outcomes at the end of a 16-week wild blueberry intervention and 16-week control period with a matched placebo.
  Quality of life will be assessed using a 32-item questionnaire that covers multiple aspects of daily living and well-being. The questionnaire asks about physical health, emotional state, social relationships, and overall life satisfaction. By combining responses across these domains, it provides a broad picture of how individuals perceive and experience their quality of life.
Other perceivable benefits: assessment of sleep by the Pittsburgh Sleep Quality Index (PSQI) | Change in sleep characteristics at the end of a 16-week wild blueberry intervention and 16-week control period with a matched placebo.
  Sleep characteristics will be assessed using the 10-item Pittsburgh Sleep Quality Index (PSQI). This standardized questionnaire asks about different aspects of sleep over the past month, including sleep duration, quality, and disturbances. By combining the responses, the PSQI provides an overall score that reflects both subjective sleep quality and potential sleep problems
Other perceivable benefits: assessment of mood by the Affect Grid | Change in mood at the end of a 16-week wild blueberry intervention and 16-week control period with a matched placebo.
  Mood will be assessed using the Affect Grid, a simple self-report tool that measures two key dimensions of emotion: pleasure (ranging from positive to negative feelings) and arousal (ranging from calm to highly activated). Participants indicate their current state on a single-page grid, providing a quick and intuitive snapshot of their mood at that moment.
Other perceivable benefits: Assessment of Stress by the Perceived Stress Scale (PSS) | Change in outcomes at the end of a 16-week wild blueberry intervention and 16-week control period with a matched placebo.
  Stress will be assessed using the Perceived Stress Scale (PSS), a widely used questionnaire that asks about feelings and thoughts during the past month. The PSS captures how unpredictable, uncontrollable, and overloaded participants perceive their lives to be. Higher scores indicate greater levels of perceived stress, providing a useful measure of everyday psychological strain.
Weight | At all test days (week 0, 8, 16, 24, 32, 40).
  Weight will be determined in kilograms.
Length | At all test days (week 0, 8, 16, 24, 32, 40).
  Length will be determined in meters.
Waist circumference | At all test days (week 0, 8, 16, 24, 32, 40).
  Waist circumference in centimeters.
Hip circumference | At all test days (week 0, 8, 16, 24, 32, 40).
  Hip circumference in centimeters.
Assessment of food intake by Food Frequency Questionnaire (FFQ) | Change in food intake at the end of a 16-week wild blueberry intervention and 16-week control period with a matched placebo.
  Food intake will be assessed using the Food Frequency Questionnaire (FFQ), a standardized dietary survey that asks participants how often they consume a wide range of foods and beverages in the past month. This method provides an overview of habitual dietary patterns, nutrient intake, and overall diet quality, making it a useful tool for linking nutrition with health outcomes.
Assessment of cerebral perfusion by Transcranial Doppler Ultrasound (TCD) | Change in cerebral perfusion by TCD will be measured during baseline and at the end of 16-week intervention (wild blueberry) or placebo period.
  Cerebral perfusion will be assessed using Transcranial Doppler ultrasound, a non-invasive method that measures blood flow in the middle cerebral artery. During the procedure, continuous blood flow velocity (CBFv) is recorded through the skull using ultrasound waves. This approach provides valuable information about the cerebrovascular health and function.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Departement of Nutrition and Movement Sciences, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wolters FJ, Zonneveld HI, Hofman A, van der Lugt A, Koudstaal PJ, Vernooij MW, Ikram MA; Heart-Brain Connection Collaborative Research Group. Cerebral Perfusion and the Risk of Dementia: A Population-Based Study. Circulation. 2017 Aug 22;136(8):719-728. doi: 10.1161/CIRCULATIONAHA.117.027448. Epub 2017 Jun 6. PMID 28588075
- [Background] Ahles S, Stevens YR, Joris PJ, Vauzour D, Adam J, de Groot E, Plat J. The Effect of Long-Term Aronia melanocarpa Extract Supplementation on Cognitive Performance, Mood, and Vascular Function: A Randomized Controlled Trial in Healthy, Middle-Aged Individuals. Nutrients. 2020 Aug 17;12(8):2475. doi: 10.3390/nu12082475. PMID 32824483
- [Background] Ivanov D, Gardumi A, Haast RAM, Pfeuffer J, Poser BA, Uludag K. Comparison of 3T and 7T ASL techniques for concurrent functional perfusion and BOLD studies. Neuroimage. 2017 Aug 1;156:363-376. doi: 10.1016/j.neuroimage.2017.05.038. Epub 2017 May 19. PMID 28528845
- [Background] Kullmann S, Veit R, Peter A, Pohmann R, Scheffler K, Haring HU, Fritsche A, Preissl H, Heni M. Dose-Dependent Effects of Intranasal Insulin on Resting-State Brain Activity. J Clin Endocrinol Metab. 2018 Jan 1;103(1):253-262. doi: 10.1210/jc.2017-01976. PMID 29095982
- [Background] Alsop DC, Detre JA, Golay X, Gunther M, Hendrikse J, Hernandez-Garcia L, Lu H, MacIntosh BJ, Parkes LM, Smits M, van Osch MJ, Wang DJ, Wong EC, Zaharchuk G. Recommended implementation of arterial spin-labeled perfusion MRI for clinical applications: A consensus of the ISMRM perfusion study group and the European consortium for ASL in dementia. Magn Reson Med. 2015 Jan;73(1):102-16. doi: 10.1002/mrm.25197. Epub 2014 Apr 8. PMID 24715426
- [Background] Azari H, Morovati A, Pourghassem Gargari B, Sarbakhsh P. Beneficial effects of blueberry supplementation on the components of metabolic syndrome: a systematic review and meta-analysis. Food Funct. 2022 May 10;13(9):4875-4900. doi: 10.1039/d1fo03715c. PMID 35445669
- [Background] Joris PJ, Plat J, Bakker SJ, Mensink RP. Long-term magnesium supplementation improves arterial stiffness in overweight and obese adults: results of a randomized, double-blind, placebo-controlled intervention trial. Am J Clin Nutr. 2016 May;103(5):1260-6. doi: 10.3945/ajcn.116.131466. Epub 2016 Apr 6. PMID 27053384
- [Background] Joris PJ, Plat J, Kusters YH, Houben AJ, Stehouwer CD, Schalkwijk CG, Mensink RP. Diet-induced weight loss improves not only cardiometabolic risk markers but also markers of vascular function: a randomized controlled trial in abdominally obese men. Am J Clin Nutr. 2017 Jan;105(1):23-31. doi: 10.3945/ajcn.116.143552. Epub 2016 Nov 23. PMID 27881395
- [Background] Nijssen KMR, Mensink RP, Plat J, Joris PJ. Longer-term mixed nut consumption improves brain vascular function and memory: A randomized, controlled crossover trial in older adults. Clin Nutr. 2023 Jul;42(7):1067-1075. doi: 10.1016/j.clnu.2023.05.025. Epub 2023 Jun 3. PMID 37296019
- [Background] Tischmann L, Adam TC, Mensink RP, Joris PJ. Longer-term soy nut consumption improves vascular function and cardiometabolic risk markers in older adults: Results of a randomized, controlled cross-over trial. Clin Nutr. 2022 May;41(5):1052-1058. doi: 10.1016/j.clnu.2022.03.014. Epub 2022 Mar 14. PMID 35395555
- [Background] Nijssen KM, Mensink RP, Plat J, Ivanov D, Preissl H, Joris PJ. Mixed nut consumption improves brain insulin sensitivity: a randomized, single-blinded, controlled, crossover trial in older adults with overweight or obesity. Am J Clin Nutr. 2024 Feb;119(2):314-323. doi: 10.1016/j.ajcnut.2023.12.010. Epub 2023 Dec 20. PMID 38128733
- [Background] Kleinloog JPD, Mensink RP, Smeets ETHC, Ivanov D, Joris PJ. Acute inorganic nitrate intake increases regional insulin action in the brain: Results of a double-blind, randomized, controlled cross-over trial with abdominally obese men. Neuroimage Clin. 2022;35:103115. doi: 10.1016/j.nicl.2022.103115. Epub 2022 Jul 14. PMID 35843050
- [Background] Nijssen KMR, Mensink RP, Joris PJ. Effects of Intranasal Insulin Administration on Cerebral Blood Flow and Cognitive Performance in Adults: A Systematic Review of Randomized, Placebo-Controlled Intervention Studies. Neuroendocrinology. 2023;113(1):1-13. doi: 10.1159/000526717. Epub 2022 Aug 24. PMID 36219990
- [Background] Kleinloog JPD, Tischmann L, Mensink RP, Adam TC, Joris PJ. Longer-term soy nut consumption improves cerebral blood flow and psychomotor speed: results of a randomized, controlled crossover trial in older men and women. Am J Clin Nutr. 2021 Dec 1;114(6):2097-2106. doi: 10.1093/ajcn/nqab289. PMID 34510189
- [Background] Rees A, Dodd GF, Spencer JPE. The Effects of Flavonoids on Cardiovascular Health: A Review of Human Intervention Trials and Implications for Cerebrovascular Function. Nutrients. 2018 Dec 1;10(12):1852. doi: 10.3390/nu10121852. PMID 30513729
- [Background] Wood E, Hein S, Mesnage R, Fernandes F, Abhayaratne N, Xu Y, Zhang Z, Bell L, Williams C, Rodriguez-Mateos A. Wild blueberry (poly)phenols can improve vascular function and cognitive performance in healthy older individuals: a double-blind randomized controlled trial. Am J Clin Nutr. 2023 Jun;117(6):1306-1319. doi: 10.1016/j.ajcnut.2023.03.017. Epub 2023 Mar 25. PMID 36972800
- [Background] Ahles S, Joris PJ, Plat J. Effects of Berry Anthocyanins on Cognitive Performance, Vascular Function and Cardiometabolic Risk Markers: A Systematic Review of Randomized Placebo-Controlled Intervention Studies in Humans. Int J Mol Sci. 2021 Jun 17;22(12):6482. doi: 10.3390/ijms22126482. PMID 34204250
- [Background] Snyder HM, Corriveau RA, Craft S, Faber JE, Greenberg SM, Knopman D, Lamb BT, Montine TJ, Nedergaard M, Schaffer CB, Schneider JA, Wellington C, Wilcock DM, Zipfel GJ, Zlokovic B, Bain LJ, Bosetti F, Galis ZS, Koroshetz W, Carrillo MC. Vascular contributions to cognitive impairment and dementia including Alzheimer's disease. Alzheimers Dement. 2015 Jun;11(6):710-7. doi: 10.1016/j.jalz.2014.10.008. Epub 2014 Dec 12. PMID 25510382
- [Background] Joris PJ, Mensink RP, Adam TC, Liu TT. Cerebral Blood Flow Measurements in Adults: A Review on the Effects of Dietary Factors and Exercise. Nutrients. 2018 Apr 25;10(5):530. doi: 10.3390/nu10050530. PMID 29693564
- [Background] Baker LD, Cross DJ, Minoshima S, Belongia D, Watson GS, Craft S. Insulin resistance and Alzheimer-like reductions in regional cerebral glucose metabolism for cognitively normal adults with prediabetes or early type 2 diabetes. Arch Neurol. 2011 Jan;68(1):51-7. doi: 10.1001/archneurol.2010.225. Epub 2010 Sep 13. PMID 20837822
- [Background] Kullmann S, Heni M, Hallschmid M, Fritsche A, Preissl H, Haring HU. Brain Insulin Resistance at the Crossroads of Metabolic and Cognitive Disorders in Humans. Physiol Rev. 2016 Oct;96(4):1169-209. doi: 10.1152/physrev.00032.2015. Epub 2016 Aug 3. PMID 27489306
- [Background] Craft S. The role of metabolic disorders in Alzheimer disease and vascular dementia: two roads converged. Arch Neurol. 2009 Mar;66(3):300-5. doi: 10.1001/archneurol.2009.27. PMID 19273747
- [Background] Neergaard JS, Dragsbaek K, Christiansen C, Nielsen HB, Brix S, Karsdal MA, Henriksen K. Metabolic Syndrome, Insulin Resistance, and Cognitive Dysfunction: Does Your Metabolic Profile Affect Your Brain? Diabetes. 2017 Jul;66(7):1957-1963. doi: 10.2337/db16-1444. Epub 2017 Apr 7. PMID 28389469
- [Background] van der Flier WM, Skoog I, Schneider JA, Pantoni L, Mok V, Chen CLH, Scheltens P. Vascular cognitive impairment. Nat Rev Dis Primers. 2018 Feb 15;4:18003. doi: 10.1038/nrdp.2018.3. PMID 29446769
- [Background] Biessels GJ, Deary IJ, Ryan CM. Cognition and diabetes: a lifespan perspective. Lancet Neurol. 2008 Feb;7(2):184-90. doi: 10.1016/S1474-4422(08)70021-8. PMID 18207116
- [Background] Gorelick PB, Scuteri A, Black SE, Decarli C, Greenberg SM, Iadecola C, Launer LJ, Laurent S, Lopez OL, Nyenhuis D, Petersen RC, Schneider JA, Tzourio C, Arnett DK, Bennett DA, Chui HC, Higashida RT, Lindquist R, Nilsson PM, Roman GC, Sellke FW, Seshadri S; American Heart Association Stroke Council, Council on Epidemiology and Prevention, Council on Cardiovascular Nursing, Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Vascular contributions to cognitive impairment and dementia: a statement for healthcare professionals from the american heart association/american stroke association. Stroke. 2011 Sep;42(9):2672-713. doi: 10.1161/STR.0b013e3182299496. Epub 2011 Jul 21. PMID 21778438
- [Background] Arnold SE, Arvanitakis Z, Macauley-Rambach SL, Koenig AM, Wang HY, Ahima RS, Craft S, Gandy S, Buettner C, Stoeckel LE, Holtzman DM, Nathan DM. Brain insulin resistance in type 2 diabetes and Alzheimer disease: concepts and conundrums. Nat Rev Neurol. 2018 Mar;14(3):168-181. doi: 10.1038/nrneurol.2017.185. Epub 2018 Jan 29. PMID 29377010